CLINICAL TRIAL: NCT06122974
Title: A RanDomized Controlled Trial of the Drug Eluting TEmporary Spur StEnt System vs PERcutaneous Balloon Angioplasty for the TReatment of CriTical Limb Ischemia
Brief Title: Drug Eluting Temporary Spur Stent System vs Percutaneous Balloon Angioplasty for the Treatment of Critical Limb Ischemia
Acronym: DEEPER RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ReFlow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CP-006
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Intervention Model Description: Phase A will enroll 20 subjects and evaluate 30-day safety data
  Phase B will enroll 345 to 518 subjects. Subjects from Phase A will be rolled into Phase B.
Who Masked: Participant
Masking Description: Subject will be blinded from their treatment assignment through the 12-month follow-up visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Study Device (Other): Subjects randomized to the Drug Eluting Temporary Spur Stent System
  Interventions: Device: Drug Eluting Temporary Spur Stent System
- Control (Other): Subjects randomized to the PTA
  Interventions: Device: Percutaneous Transluminal Balloon Angioplasty

INTERVENTIONS:
Device: Drug Eluting Temporary Spur Stent System — The Spur Stent consists of a sirolimus coated stent and balloon that is retrievable after delivery of the sirolimus formulation.
  Arms: Study Device
Device: Percutaneous Transluminal Balloon Angioplasty — A balloon catheter is inserted across a lesion and inflated to fracture and compress the plaque, creating a larger lumen and improved blood flow through the artery.
  Arms: Control

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of the Drug Eluting Temporary Spur Stent System compared to PTA.

The Drug Eluting Temporary Spur Stent System is intended for use as a primary treatment in the infrapopliteal arteries for the treatment of de novo or restenotic lesions.

DETAILED DESCRIPTION:
This is a randomized controlled trial evaluating the safety and efficacy of the Drug Eluting Temporary Spur Stent System (Spur) compared to percutaneous transluminal balloon angioplasty (PTA). The trial will be conducted in two phases.

Phase A is a prospective, multi-center, 1:1 randomized dual arm study of 20 subjects, evaluating the short-term safety of the Drug Eluting Temporary Spur Stent System compared to PTA to treat lesions in infrapopliteal arteries in subjects with critical limb ischemia (CLI). Thirty (30) day data from Subjects in Phase A will be evaluated by an independent Data Safety Monitoring Board (DSMB) and submitted to the Food and Drug Administration (FDA) for review. Phase A subjects will be rolled into Phase B.

Phase B is a prospective, multicenter, 1:1 randomized dual arm study of no less than 345 and up to 518 subjects, evaluating the safety and efficacy of the Drug Eluting Temporary Spur Stent System compared to PTA to treat lesions in infrapopliteal arteries in subjects with CLI.

ELIGIBILITY:
Inclusion Criteria:

Pre-Procedure Inclusion Criteria:

1. Subject willing and able to provide informed consent and able to comply with the study protocol and follow up. Subjects who are unable to sign due to a physical limitation may have a Legally Authorized Representative (LAR), including a family member, sign on their behalf.
2. Life expectancy greater than 1 year in the investigator's opinion.
3. Subject is greater than 18 years of age.
4. Subjects must have chronic (greater than 14 days) symptoms of limb ischemia, determined by clinical symptoms of Rutherford class 4-5, rest pain (R4), and/or minor tissue loss (R5), that in the opinion of the investigator are not amenable to conservative medical therapy and require endovascular intervention for alleviation of symptoms and tissue preservation.
5. For subjects with bilateral disease, planned treatment of the contralateral limb must either be performed greater than or equal to 7 days prior to the index procedure or greater than or equal to 30 days following the index procedure.

Angiographic Inclusion Criteria:

1. Stenotic, restenotic, or occlusive lesions with greater than or equal to 70% stenosis located in the infrapopliteal vessels, with target lesion that can be successfully crossed with a guidewire via the true lumen.
2. Iliac, Superficial Femoral Artery (SFA) and popliteal inflow lesions can be treated using standard of care during the index procedure

   Note:
   1. Inflow lesions treated intraprocedure must be treated first, prior to consideration of treatment of infrapopliteal lesions.
   2. Treatment of in-stent restenosis in inflow treatment is permitted, provided that stents are not severely fractured or otherwise compromised.
   3. Distal embolic protection is strongly encouraged in cases where atherectomy is used.
   4. Inflow lesions must have a healthy vessel segment of greater than 30 mm between the study lesion and the treated segment, defined as less than 50% stenosis without aneurysmal segments.
   5. Inflow treatment must be successful, prior to treatment of the target lesion, resulting in stenosis less than or equal to 30%, without resulting flow limiting (Type D or greater) dissection, thrombus, or aneurysm by angiography prior to randomization.
3. Target vessel reconstitutes at or above the ankle, with the target treated segment ending at least 10 mm above the ankle joint.

   Note:
   1. If the anterior tibial or posterior tibial arteries are treated, there must be inline flow to the foot.
   2. If the peroneal artery is treated, there must be at least one collateral supplying the foot.
   3. In all cases, patent runoff (no lesions with greater than 50% stenosis) must be present via the dorsalis pedis and/or plantar arteries.
4. Target lesion must be located in the tibial arteries. If vessel sizing remains appropriate, treatment may extend into the distal popliteal (P3) segment.
5. Target vessel reference diameter is measured to be greater than or equal to 2.5 and less than or equal to 4.25 mm in diameter assessed by one of the following methods after successful completion of guidewire crossing of the lesion site (visual estimate permitted):

   1. Intravascular Ultrasound (IVUS)
   2. Quantitative Vascular Angiography (QVA)
   3. Visual Estimate
6. Target lesion length must be less than or equal to 210 mm cumulatively. Tandem lesions that are less than or equal to 4 cm should be treated as one lesion. Multiple discrete lesions may be treated provided cumulative length is less than or equal to 210 mm.
7. Only one limb and one vessel may be enrolled per subject. If the investigator feels that multiple infrapopliteal vessels must be treated during the index procedure, a standard practice treatment may be performed in the non-target infrapopliteal vessel(s). This should be prior to randomization of and treatment of the target vessel whenever possible.

   Note:
   1. Distal embolic protection is strongly recommended in cases using atherectomy.
   2. Treatment of the target vessel/lesion may be performed only if treatment of the non-target vessel(s)/lesion(s) does not result in a complication which may compromise the outflow of the target lesion or result in a major adverse limb event.
   3. Treatment of non-target lesions must be parallel to, and not contiguous with, the target lesion.
8. Retrograde access (in the infrapopliteal arteries) is permitted for lesion crossing; however, the randomized treatment must be deployed from antegrade (above the knee, either ipsilateral or contralateral) access.

Exclusion Criteria:

Pre-procedure Exclusion Criteria:

1. Subject unwilling or unlikely to comply with the 5-year duration of the study in the opinion of the investigator.
2. Subject is pregnant or planning to become pregnant during the course of the trial.
3. Subject is breastfeeding or planning to breastfeed during the course of the trial.
4. Subject has an active systemic infection that is not controlled at the time of the procedure, including septicemia or bacteremia.
5. Subject has osteomyelitis proximal to the phalanges of the target foot. Osteomyelitis in the digit(s) of the target foot is permitted.
6. Wounds in the target limb must be confined to the foot below the ankle.
7. Heel wounds on the target foot are excluded; wounds on the plantar surface of the hindfoot are permitted.
8. Planned major (above the ankle) amputation of the target limb. A planned or previous minor (transmetatarsal amputation or digit amputation) amputation) is permitted.
9. Myocardial infarction (MI) or stroke within 90 days of the index procedure.
10. Symptomatic acute heart failure New York Heart Association (NYHA) class III or greater.
11. Impaired renal function (estimated Glomerular Filtration Rate (eGFR) less than or equal to 25 mL/min) within 30 days of procedure or end stage renal disease on dialysis.
12. Subject with vasculitis or uncontrolled clotting disorder that may preclude patient to thrombotic events.
13. Inability to tolerate dual antiplatelet and/or anticoagulation therapy, including a history of severe bleeding or coagulopathy.
14. Known allergies or sensitivities to heparin, antiplatelet drugs, other anticoagulant therapies which could not be substituted, drug balloon coatings and their excipients, including, but not limited to, paclitaxel, sirolimus, or zotarolimus, or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
15. The subject is currently enrolled in another investigational device or drug trial that interferes with the study endpoints.
16. Known allergy to nitinol or nickel.
17. Bypass surgery of the target vessel. Prior bypass above the level of the infrapopliteal arteries is permitted.

Angiographic Exclusion Criteria

1. Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion. Inflow must also be free of unstable or flow limiting aneurysmal segments.
2. Fractured or otherwise compromised stents or dissection repair devices in the target vessel or inflow vessel.
3. In-stent restenosis in the target vessel, including restenosis of dissection repair devices.
4. Previous treatment of the target vessel less than or equal to 90 days prior to index procedure.
5. Angiographic evidence of thrombus within target limb.
6. Extremely severe calcification that, in the investigator's opinion, would not be amenable to PTA.
7. Flow-limiting dissection incurred during lesion crossing
8. Significant (greater than or equal to 70%) stenosis of inflow arteries or unsuccessful treatment of inflow lesions.
9. Distance from access to lesion is too long for 135 cm working length of catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2032-06 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Phase A: Primary Safety Endpoint | 30 Days
  Freedom from the occurrence of major adverse limb events (MALE), and peri-operative death (POD), in Drug Eluting Temporary Spur Stent System and PTA-treated subjects through 30 days post-procedure. MALE are defined as:
  * Major amputation above the ankle
  * Major (open vascular surgery) reintervention
  * Target vessel thrombectomy or thrombolysis
Phase B: Primary Safety Endpoint | 30 Days & 6 Months
  Freedom from the occurrence of POD at 30 days, and the occurrence of MALE at 6 months.
Phase B: Primary Efficacy Endpoint | 6 Months
  Freedom from a composite endpoint of the occurrence of limb salvage and primary patency events at 6 months, defined as:
  * Clinically-driven target lesion revascularization (CD-TLR).
  * Above the ankle amputation in the index limb, in the presence of a totally occluded target vessel.
  * 100% total occlusion of target lesion in Spur and PTA-treated subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood Razavi, MD, Principal Investigator — Providence Hospital St. Joseph; S. Jay Mathews, MD, Principal Investigator — Manatee Memorial Hospital

IPD SHARING:
Plan to Share IPD: No